CLINICAL TRIAL: NCT00632099
Title: Progesterone Treatment for Cocaine-dependent Women: A Pilot Study
Acronym: PROG
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #5568; R01DA022218 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2008-03-06; First posted 2008-03-10 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Cocaine Dependence
Keywords: cocaine; treatment; progesterone
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): matched placebo
  Interventions: Drug: Placebo
- Oral micronized progesterone (Experimental): Oral micronized progesterone (up to 400 mg/day)
  Interventions: Drug: Oral micronized progesterone

INTERVENTIONS:
Drug: Oral micronized progesterone — Oral micronized progesterone (up to 400 mg/day), suspended in olive oil
  Other Names: Progesterone
  Arms: Oral micronized progesterone
Drug: Placebo — matched placebo
  Arms: Placebo

SUMMARY:
The purpose of this pilot treatment trial is to evaluate the efficacy of oral micronized PROG in cocaine-dependent women. Since we have shown (Evans & Foltin, 2006) that oral micronized PROG attenuates the positive subjective effects of smoked cocaine in females, but not in males, and we have preliminary data indicating that oral micronized PROG also reduces smoked cocaine self-administration in the laboratory, PROG appears to be an ideal potential candidate medication to evaluate in cocaine-dependent women. Prior to randomization to treatment, women will reside inpatient for one week to ensure cocaine abstinence since one of the primary outcome measures will be time to cocaine relapse.

DETAILED DESCRIPTION:
Primary Aims: The primary aims will be directed at treatment efficacy. Relatively unique to cocaine treatment trials, one of the principal outcome measures will be time to cocaine relapse. We hypothesize that maintenance on PROG will increase the time to cocaine relapse compared to maintenance on placebo (PBO). Another cocaine-related efficacy endpoint will be the proportion of patients who achieve at least 2 consecutive weeks of cocaine abstinence (based on urine toxicology results) during the double-blind treatment phase. Lastly, the proportion of cocaine-negative urines collected throughout the treatment trial will be measured. We hypothesize that women in the PROG group will show a greater reduction in cocaine use compared to those in the PBO group.

Secondary Aims: 1) Determine if response to laboratory stressors will predict treatment outcome. We hypothesize that those women with the greatest stress response will do worse in treatment and that maintenance on PROG will reduce stress/anxiety and thereby improve treatment outcome. 2) Determine if treatment retention is better in the PROG group compared to the PBO group and determine if maintenance on PROG improves overall functioning compared to maintenance on PBO based on the Clinical Global Inventory (CGI). We hypothesize that women in the PROG group will have better treatment retention and improvement in CGI scores compared to women in the PBO group.

Tertiary Aims: To conduct exploratory analyses to determine whether 1) trauma history is related to treatment outcomes and 2) improvements in treatment outcome measures are related to decreases in HIV high-risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women between the ages of 18-60 who meet criteria for current cocaine dependence (DSM-IV-TR). Volunteers may meet criteria for abuse or dependence on nicotine, marijuana or alcohol, as long as the dependence is secondary to cocaine dependence and does not require any medical intervention (see additional exclusions for alcohol dependence below).

  2. Use cocaine by the smoked or intranasal route at least four days in the past month, with at least weekly cocaine use.

  3. Women with regular menstrual cycles (24-45 days) who are not pregnant, based on the results of a blood pregnancy test drawn at the time of screening. They must agree to use a barrier method of contraception with proven efficacy and agree not to become pregnant during the study. To confirm this, urine pregnancy tests will be conducted weekly.

  4. Women must be capable of giving informed consent and capable of complying with study procedures.

Exclusion Criteria:

* 1. Meets DSM-IV-TR criteria for bipolar disorder, Schizophrenia, or any psychotic disorder other than transient psychosis due to drug abuse.

  2. Individuals with any current Axis I psychiatric disorder as defined by DSM-IV-TR supported by the SCID-I/P that in the investigator's judgment are unstable or would be disrupted by study medication. Disorders that are stable on psychotherapy or pharmacotherapy will not be exclusionary. Individuals will be permitted to take prescribed zolpidem and zaleplon or other medications for insomnia if there is no evidence of dependence on these substances.

  3. Individuals with current major depressive disorder.

  4. Individuals physiologically dependent on any other drugs (excluding nicotine or cannabis) that require medical intervention will be excluded and referred for treatment. Individuals with severe alcohol dependence , even without physiological dependence, or with any known alcohol-related diseases will also be excluded.

  5. Females who have any of the following medical contraindications: undiagnosed abnormal genital bleeding, known or suspected history of breast or genital cancer, active deep vein thrombosis, pulmonary embolism, or history of these conditions, active or recent (within last year) arterial thromboembolic diseases (e.g., stroke, myocardial infarction), liver dysfunction.

  6. Females who are cognitively impaired or have a chronic organic mental disorder.

  7. Individuals with current suicidal risk.

  8. Individuals with coronary vascular disease as indicated by history or suspected by abnormal ECG or history of cardiac symptoms.

  9. Unstable physical disorders which might make participation hazardous such as uncontrolled hypertension (Blood pressure > 150/ 90, or Heart Rate > 100 when sitting quietly), acute hepatitis (patients with chronic mildly elevated transaminases < 3x upper limit of normal are acceptable), or uncontrolled diabetes.

  10. Individuals with a history of seizures.

  11. Women who are pregnant or nursing.

  12. Individuals who are legally mandated (e.g., to avoid incarceration, monetary or other penalties, etc.) to participate in substance abuse treatment program.

  13. Females with a known or suspected hypersensitivity to oral micronized progesterone.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2008-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Evans, PhD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Oliva A, Reed SC, Brooks DJ, Levin FR, Evans SM. Safety and tolerability of progesterone treatment for women with cocaine use disorder: a pilot treatment trial. Am J Drug Alcohol Abuse. 2022 Sep 3;48(5):586-595. doi: 10.1080/00952990.2022.2114004. Epub 2022 Sep 12. PMID 36095308
- See also: Substance Treatment and Research Service of Columbia University — http://www.stars.columbia.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Matched Placebo: matched placebo
  Placebo: matched placebo
Period: Overall Study
Arm/Group | Matched Placebo | Oral Micronized Progesterone
Started | 10 | 11
Completed | 7 | 8
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Matched Placebo | Oral Micronized Progesterone | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (9) | 45 (8) | 43 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 5 | 4 | 9
  Black | 4 | 5 | 9
  Hispanic | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Abstinence Based on Urine Toxicology Results
Description: Percentage of patients cocaine abstinent during last 3 weeks of the study (weeks 7-9)
Time Frame: during last 3 weeks of the trial
Measure: Number; unit: participants
Arm/Group | Matched Placebo | Oral Micronized Progesterone
Number analyzed (Participants) | 10 | 11
participants | 1 | 3
Statistical Analysis 1: Comparison: Matched Placebo vs Oral Micronized Progesterone; Test type: Superiority or Other; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: 10 weeks of study participation
Arm/Group | Matched Placebo | Oral Micronized Progesterone
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/11
Other Adverse Events (participants affected / at risk) | 8/10 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matched Placebo (N=10) | Oral Micronized Progesterone (N=11)
Uveitis (Eye disorders) | 0 (0) | 1 (1) — Patient experienced pain and floater and was diagnosed with uveitis. The patient was followed by her ophthalmologist and two weeks later and had outpatient laser surgery for retinal detachment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matched Placebo (N=10) | Oral Micronized Progesterone (N=11)
abdominal pain/cramps (Reproductive system and breast disorders) | 1 (1) | 3 (3)
breast tenderness (Reproductive system and breast disorders) | 4 (4) | 2 (2)
headache (General disorders) | 6 (6) | 4 (4)
fatigue (General disorders) | 5 (5) | 3 (3)
chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 2 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
dizziness (General disorders) | 2 (2) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
swollen hands (General disorders) | 1 (1) | 0 (0)
increased libido (General disorders) | 0 (0) | 1 (1)
hot flashes (General disorders) | 0 (0) | 1 (1)
irritability (Psychiatric disorders) | 1 (1) | 1 (1)
eye discomfort (Eye disorders) | 0 (0) | 2 (2)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
increased appetite (Gastrointestinal disorders) | 2 (2) | 0 (0)
dry mouth (General disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Given the limited sample size, it was not possible to adequately determine whether OM-PROG may be an effective treatment for cocaine-dependence in women, but it was well tolerated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes